CLINICAL TRIAL: NCT06933667
Title: Kimel Family Centre for Brain Health and Wellness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: #23-26
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Prevention; Dementia
Keywords: personalized dementia prevention; lifestyle factors
MeSH Terms: conditions — Dementia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are encouraged to sign up for programs that address their specific cluster of modifiable dementia risk factors in five domains: physical activity, brain-healthy eating, cognitive engagement, social connections, and mental wellbeing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Physical Activity (Active Comparator): Participants are encouraged to work up to the Canadian Guidelines of 150 minutes a week of moderate to vigorous activity and to focus on balance and stretching.
  Interventions: Behavioral: Physical Activity
- Brain-healthy Eating (Active Comparator): Participants are recommended to take five required courses about the CCNA Brain Health Food Guide, then take additional courses of their choice.
  Interventions: Behavioral: Brain-healthy Eating
- Cognitive Engagement (Active Comparator): Participants are encouraged to participate in at least one hour of cognitively engaging programs.
  Interventions: Behavioral: Cognitive Engagement
- Social Connections (Active Comparator): All programs, regardless of type, encourage social connections, through ice-breakers, peer mentoring, and time to chat before and after classes.
  Interventions: Behavioral: Social Connections
- Mental Wellbeing (Active Comparator): Participants are encouraged to participate in at least one hour of programming focused on mental wellbeing (e.g., meditation, relaxation).
  Interventions: Behavioral: Mental Wellbeing

INTERVENTIONS:
Behavioral: Physical Activity — Participants can chose (with input from a kinesiologist as required) from courses of varying intensity in our gym, warm water pool, or classrooms.
  Arms: Physical Activity
Behavioral: Brain-healthy Eating — Participants take five foundational courses: Brain-healthy eating, Healthy protein choices, Colour your diet: Maximize the benefits of fruits and vegetables; Interpreting nutrition facts labels; and Salt and sugar: How much is too much? They are also encouraged to take additional nutrition programs.
  Arms: Brain-healthy Eating
Behavioral: Cognitive Engagement — Participants can sign up for any lecture, discussion group, book club, creative arts program, etc. linked to the Cognitive Engagement risk factor.
  Arms: Cognitive Engagement
Behavioral: Social Connections — Social Connections are baked into all other programming. Our instructors are trained in how to foster connections among participants, through peer coaching, ice-breakers, etc., and are asked to leave some time at the beginning and end of programs for participants to chat. We also hold special social events such as game nights.
  Arms: Social Connections
Behavioral: Mental Wellbeing — Participants are encouraged to enroll in one a week of relevant programming (e.g., meditation, relaxation).
  Arms: Mental Wellbeing

SUMMARY:
Participants (n=450; aged 50+; without a diagnosis of dementia; sufficiently fluent in English to complete the assessments and engage in programming) receive a comprehensive dementia risk assessment, including nonmodifiable and modifiable risk factors, from which they receive a Personalized Dementia Risk Report and Program Strategy, indicating their health conditions increasing and their risk level in five modifiable risk domains: physical activity, brain- healthy eating, cognitive engagement, social connections, and mental wellbeing. Equipped with this information, participants enroll in programs within the Centre to address their risk factors. Changes to their dementia risk, cognition, and Personalized Program Strategy are communicated through re-assessments of risk factors every six months (risk and cognition) and every year (comprehensive assessment).

DETAILED DESCRIPTION:
Participants (n=450; aged 50+; without a diagnosis of dementia; sufficiently fluent in English to complete the assessments and engage in programming) complete a baseline assessment consisting of three parts. A biosample session in which blood is drawn to measure HbA1c, cholesterols, thyroid levels, c-reactive protein, interleukin-6, homocysteine, and BDNF, and a saliva sample is provided to provide a polygenic risk score for AD. A questionnaire session is completed on a tablet or from home asks about demographics, health conditions, and five targeted modifiable factors: physical activity, brain-healthy eating, cognitive engagement, social connections, and mental wellbeing. A clinical session measures vitals, sensory function, frailty markers (grip strength, DXA, ultrasound of right quadriceps muscle), dual-task gait, and cognition (MoCA and Cogniciti's Brain Health Assessment). From that assessment, participants receive a Personalized Dementia Risk Report and Program Strategy, outlining conditions that are known to increase dementia risk, with resources provided on how to get them addressed, as well as their risk level in the five targeted domains. Participants then take a SMART goal setting workshop to identify SMART goals addressing their dementia risk factors, and then sign up for programming in the centre to reduce their risk. After six months, their risk in the five targeted domains, cognition (Brain Health Assessment), and satisfaction are re-assessed, and every year, most of the baseline assessment is repeated. We expect that this personalized approach will result in reductions in risk in the five targeted domains within the first six months, improvements in health factors within the first year, and improvements in cognition within two years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older
* Sufficiently fluent in English to complete the assessments and participate in programming.

Exclusion Criteria:

* Diagnosis of dementia.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | Every six months over two years.
  Hours of moderate-to-vigorous physical activity a week, as determined by the CHAMPS (0 - 168, with higher scores indicating greater activity).
Cognition | We expect to see this at the two year mark.
  We expect cognition to be maintained or improved, as assessed by Cogniciti's Brain Health Assessment, to the extent that participants adhere to their Personalized Program Strategy.
Brain-Healthy Eating | Every six months over two years.
  Brain-healthy eating as assessed by the Brain Health Food Guide derived Eating Pattern Self-Assessment (range 0 - 15, with higher scores indicating greater adherence to the Brain Health Food Guide).
Cognitive Engagement | Every six months over two years.
  Amount of engagement in higher-order cognitively engaging activities, as assessed by the Higher Cognition subscale of the Florida Cognitive Activities Scale (range 0-40, with higher scores indicated greater engagement).
Social Connections | Every six months over two years.
  Degree of loneliness as assessed by the UCLA Loneliness Scale (Version 3; range = 0-80, where higher scores indicate greater loneliness).
Mental Wellbeing | Every six months over two years.
  A composite of depression, anxiety, and (dis)stress from the Depression, Anxiety, and Stress Scale-21 (DASS-21), as well as perceived stress from the Perceived Stress Scale (with each subscale converted to a percentage of maximum and summed; range: 0 - 400).
Diastolic Blood Pressure | Every year over two years.
  Diastolic Blood Pressure, which lower numbers indicated better blood pressure.
Systolic Blood Pressure | Every year over two years.
  Systolic Blood Pressure, where lower numbers indicate better blood pressure
Percent body fat | Every year over two years.
  Percent body fat as determined by dual-energy X-ray absorptiometry (DXA), where lower numbers indicate less body fat.
Low density lipoprotein | Every year over two years.
  Low density lipoprotein, assessed via blood draw, where lower numbers indicate less cholesterol.
C-reactive protein | Every year over two years.
  C-reactive protein, assessed via blood draw, where lower numbers indicate less inflammation.
Interleukin-6 | Every year over two years.
  Interleukin-6, assessed via blood draw, where lower numbers indicate less inflammation.
HbA1c | Every year over two years.
  Hemoglobin A1C (HbA1c), measured through blood draw, where lower numbers indicate less blood sugar.
Cognition | Every six months over two years.
  Cognition, assessed as an age- and sex-adjusted percentile on the Brain Health Assessment (an online cognitive assessment of episodic memory, working memory, and executive functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole D. Anderson, PhD, CPsych, Principal Investigator — Baycrest; Howard Chertkow, MD, Principal Investigator — Baycrest
Locations (1):
- Baycrest, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participants are asked during consent if they consent to Open Science (as per Canadian TriCouncil Guidelines). For those who do, we will deposit the data on the Open Science Framework within three years of study completion. Data requests can also be made prior to this point by completing a Data Request Form (available from the PIs).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The study protocol has been published (http://dx.doi.org/10.14283/jpad.2024.98); the only exception is that due to funding, we are not currently including the episodic future simulation aspect of that report. That also describes our statistical analysis plan. The analytic code will be posted on OSF with the primary paper(s).
Access Criteria: When it is on OSF, anyone can access it.
URL: https://osf.io

REFERENCES:
- [Background] Anderson ND, D'Amico D, Rotenberg S, Addis DR, Gillen J, Moore D, Furlano JA, Tan B, Binns M, Santarossa M, Chertkow H. Validation of a Community-Based Approach Toward Personalized Dementia Risk Reduction: The Kimel Family Centre for Brain Health and Wellness. J Prev Alzheimers Dis. 2024;11(5):1455-1466. doi: 10.14283/jpad.2024.98. PMID 39350393
- See also: Related Info — https://kimelcentre.baycrest.org